CLINICAL TRIAL: NCT02711423
Title: A Single-Center, Randomized, Investigator/Subject-Blind Single-Ascending Dose, Placebo-Controlled, Parallel Study to Investigate the Safety, Tolerability, and Pharmacokinetics of Gantenerumab Following SC Administration in Healthy Subjects
Brief Title: A Single-Dose Study to Investigate the Safety, Tolerability, and Pharmacokinetics (PK) of Gantenerumab Following Subcutaneous (SC) Administration in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP30042; 2015-005132-17 (EudraCT Number)
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — gantenerumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part I (Dose Escalation): Gantenerumab (Experimental): Participants will receive a single SC dose of gantenerumab on Day 1.
  Interventions: Drug: Gantenerumab
- Part I (Dose Escalation): Placebo (Placebo Comparator): Participants will receive a single SC dose of matching placebo on Day 1.
  Interventions: Drug: Placebo
- Part II (PK Extension): Gantenerumab (Experimental): Participants will receive a single SC dose of gantenerumab on Day 1. The dose range will be determined by safety and tolerability data collected from Part I.
  Interventions: Drug: Gantenerumab

INTERVENTIONS:
Drug: Gantenerumab — Gantenerumab will be supplied as a high-concentration liquid formulation for SC injection into the abdomen. The single dose will be administered on Day 1.
  Arms: Part I (Dose Escalation): Gantenerumab; Part II (PK Extension): Gantenerumab
Drug: Placebo — Placebo will be supplied as a matching liquid formulation for SC injection into the abdomen. The single dose will be administered on Day 1.
  Arms: Part I (Dose Escalation): Placebo

SUMMARY:
This two-part study is designed to assess the safety, tolerability, and PK of gantenerumab in healthy volunteers. Part I (dose escalation) will randomly assign participants to receive a single blinded SC dose of gantenerumab or placebo. Part II (PK extension) will randomly assign participants to receive a single open-label SC dose of ganenerumab at different dose levels according to safety assessments from Part I.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males 18 to 45 years of age, inclusive
* Body mass index (BMI) 20.0 to 32.0 kilograms per meter-squared (kg/m^2), inclusive

Exclusion Criteria:

* History of cancer or any clinically significant disease affecting one of the major organ systems
* Prior administration of gantenerumab
* Clinically significant laboratory test results
* Clinically relevant history of hypersensitivity or allergic reaction following exposure to a drug, food, or environmental agent
* Known hypersensitivity to gantenerumab or excipients of study drug formulation
* Abnormal skin condition or potentially obscuring tattoo, pigmentation, or lesion in the area intended for SC injection
* Familial history of early-onset Alzheimer's disease

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-03-31 (Actual); Primary Completion 2016-09-28 (Actual); Study Completion 2016-09-28 (Actual)

PRIMARY OUTCOMES:
Percentage of participants with adverse events (AEs) | Up to 12 weeks (from Baseline to Day 85 +/- 5 days)

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of gantenerumab | Predose (0 hours) and 1, 6, and 12 hours from single dose administration; once daily from Days 2 to 10; and once daily on Days 12, 15, 21, 29, 43, 64, and 85
Area under the plasma concentration-time curve (AUC) of gantenerumab | Predose (0 hours) and 1, 6, and 12 hours from single dose administration; once daily from Days 2 to 10; and once daily on Days 12, 15, 21, 29, 43, 64, and 85

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Bioclinica Research, Orlando, Florida, United States